CLINICAL TRIAL: NCT02940951
Title: Integrating a Quality of Life Assessment and Practice Support System in Home Care Services for Older Adults With Chronic Life-limiting Illness and Their Families
Brief Title: Quality of Life Assessment and Practice Support System in Home Care Services for Older Adults
Acronym: QPSS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Trinity Western University (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Richard Sawatzky, Professor, Trinity Western University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: FH-REB 2015-139
Record Dates: First submitted 2016-07-05; First posted 2016-10-21 (Estimated); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: Chronic Disease; Life-limiting Illness; Palliative Care
MeSH Terms: conditions — Chronic Disease

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual home care provided by clinicians (Other): Usual care provided by the home health clinicians. This may or may not include use of some standardized forms of quality of life assessment that were in place prior to the study beginning.
  Interventions: Other: Usual care
- Use of QPSS by home health clinicians (Experimental): Usual home care plus the use of the Quality of Life Assessment and Practice Support System (QPSS) to document, monitor and address the quality of life concerns of patients and family caregivers.
  Interventions: Other: QPSS; Other: Usual care

INTERVENTIONS:
Other: QPSS — Home care providers use the QPSS that includes standardized instruments for assessing patient and family caregiver quality of life in routine care. In addition to instant calculation of scores, the QPSS allows for tracking scores over time and sharing them with other registered users from that home care service.
  Other Names: Quality of Life Assessment and Practice Support System
  Arms: Use of QPSS by home health clinicians
Other: Usual care — Home healthcare services provided by nurses and, where applicable, multi-professional teams.

SUMMARY:
Older adults living with incurable and advancing life-limiting illness frequently desire to spend as much time as possible comfortably at home, rather than in hospital. They often have complex problems that not only affect their ability to function, but also their and their family caregivers' overall quality of life (QOL). Routine assessment of their perceived health care needs and their self-reported QOL is necessary to ensure that patients' and family caregivers' concerns are visible to home care clinicians so that they can be effectively monitored and addressed. These types of assessments involve asking people to respond to questions about their symptoms, their physical, psychological, social and existential/spiritual wellbeing, and their experiences with health care. Electronic information systems are increasingly used and recommended to facilitate such QOL assessments. However, there is a need for information about how such systems are best translated into practice improvements that ultimately may improve patient- and family-centred outcomes. This study is about the implementation of an innovative, electronic health care information and practice support system, the Quality of life Assessment and Practice Support System (QPSS), into routine care provided by home care services for older adults with life-limiting illnesses and their family caregivers. Eight home care sites in Canada are participating. At each site the investigators will first adapt the QPSS to the local context and develop a plan for its local implementation. Then home care staff will be asked to use it in practice and the investigators will evaluate the process of using the QPSS and its effect on patient and family caregiver quality of life, health, and satisfaction with care as well as the cost consequences of its integration into practice. The effect of its use will be studied in a randomized trial, which is the part of the study described in this registry. Patients and their family caregivers will be randomly assigned to 1) have their home care team use the QPSS in their care or 2) not to use it, instead receiving care as usual. The effect of using the QPSS will be measured using questionnaires completed by the participating patients and family caregivers every two months. If using the QPSS improves quality of life, health, or satisfaction with care, the last stage will explore how to scale up use of the QPSS in practice and its integration with existing health information systems.

DETAILED DESCRIPTION:
Older adults living with incurable and advancing life-limiting illness frequently desire to spend as much time as possible comfortably at home, rather than in hospital. They often have complex problems that not only affect their ability to function, but also their and their family caregivers' overall quality of life (QOL). Routine assessment of their perceived health care needs and their self-reported QOL is necessary to ensure that patients' and family caregivers' concerns are visible to home care clinicians so that they can be effectively monitored and addressed. These types of assessments involve asking people to respond to questions about their symptoms, their physical, psychological, social and existential/spiritual wellbeing, and their experiences with health care. Electronic information systems are increasingly used and recommended to facilitate such QOL assessments. However, there is a need for information about how such systems are best translated into practice improvements that ultimately may improve patient- and family-centred outcomes. This study will try to improve patient and family caregiver QOL while improving the efficacy of the health care system by studying the implementation of an innovative health care information system, the Quality of life Assessment and Practice Support System (QPSS), into routine care provided by home care services for older adults with life-limiting illnesses and their family caregivers.

Research aims and questions:

This integrated knowledge translation project involves working with clinicians, patients, and family caregivers to answer the following aims and research questions.

Aim 1: To examine the efficacy of the QPSS in home care for older adults who have advancing life-limiting illnesses.

• Does the routine use of the QPSS in home care improve quality of care, as indicated by patients' and family caregivers' reports of enhanced QOL and experiences with the care provided?

Aim 2: To evaluate the cost consequences of implementing the QPSS in home care.

Aim 3: To understand the process of implementing the QPSS in home care.

• How can the integration and routine use of the QPSS in the home care for older adults who have advancing life-limiting illnesses and their family caregivers be best facilitated?

Aim 4: To examine how integration of the QPSS with health information systems will meet the needs of administrators for quality improvement and accreditation.

Design:

This project will be conducted in 3 stages at 8 home care service sites:

Stage 1: The local adaptation stage will use qualitative methods (user-centered design focus groups and interviews with clinicians, managers, patients, and family caregivers) to adapt the QPSS to the unique context of each home care service site and develop site-specific protocols for its routine integration in daily practice. For evaluative purposes, this stage will also include (a) measurement of patient and family caregiver QOL and their health care experiences prior to integrating routine use of the QPSS into home care to serve as a pre-intervention comparator group (Aim 1) and (b) data collection regarding the cost of local adaptation of and training to use the QPSS (Aim 2).

Stage 2: During the evaluation stage, the investigators will (a) conduct a randomized controlled trial to evaluate the impact of using the QPSS on the QOL and care experiences of patients and their family caregivers (Aim 1); (b) conduct an economic evaluation to estimate the cost consequences of implementing the QPSS in home care (Aim 2); and (c) apply qualitative and quantitative methods to examine the process of using the QPSS in home health care (Aim 3). The investigators aim to recruit 540 patients and 540 family caregivers. Patient participants will be 55 years of age and older who are receiving ongoing home care due to advancing life-limiting illnesses. Family caregiver participants are identified as eligible and competent by the patient, or by a clinician if the patient is unable to do so, and as the person most involved in the care of a patient who meets the abovementioned eligibility criteria. No more than one caregiver per patient will be recruited. Patient and family caregiver participants must have the ability to speak English and capacity to provide informed consent.

STAGE 3: The sustainability stage will focus on (a) whether the results warrant sustained and widespread integration of the QPSS into practice, and if so, (b) how to scale this up, (c) how to further integrate the QPSS with other health information systems to facilitate use by health care administrators for continuous quality improvement and accreditation (Aim 4) and (d) dissemination of results.

The initial patient and family caregiver consent (prior to the start of stage 2) was for 12 months from start of enrollment. They were subsequently invited to continue beyond 12 months, for up to 24 months, to allow for secondary analyses of extended trajectories of the primary and secondary outcome measures.

The start and end dates and recruitment information for this registration pertains only to the randomized controlled trial in stage 2 (evaluation).

ELIGIBILITY:
Inclusion Criteria:

1. Patients:

   * >= 55 years of age
   * receiving ongoing home care because of having one or more advancing life-limiting illnesses
   * able to speak English
   * able to provide informed consent
2. Family caregivers:

   * identified as eligible and competent by the patient, or by a clinician if the patient is unable to do so, as the person most involved in the care of a patient who meets the eligibility criteria just above (#1). No more than one caregiver per patient will be recruited
   * able to speak English
   * able to provide informed consent

Exclusion criteria:

Patients who are less than 55 years old and are not identified as having one or more advancing life-limiting illnesses.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 565 (Actual)
Dates: Start 2018-03-12 (Actual); Primary Completion 2020-05-06 (Actual); Study Completion 2021-08-06 (Actual)

PRIMARY OUTCOMES:
Differences in trajectories of change between groups in McGill Quality of Life Questionnaire -Expanded [MQOL-E] Total Score | Trajectories over 12 months from start of enrollment in Stage 2 until study completion (assessments completed every two months)
  The McGill Quality of Life Questionnaire -Expanded has 20 items covering Physical, Psychological, Existential, Social, Feeling like a burden, Environment, Cognition and Quality of health care domains. The total score is the mean of the domain scores, with possible values ranging from 0 (worst possible quality of life) to 10 (best possible quality of life).
Differences in trajectories of change between groups in Quality of Life in Life-Threatening Illness- Family (QOLLTI-F) (version 3) Total Score | Trajectories over 12 months from start of enrollment in Stage 2 until study completion (assessments completed every two months))
  Quality of Life in Life-Threatening Illness- Family (version 3) includes 16 items measuring 7 domains that contribute to quality of life: Environment; Patient Condition; Caregiver's Own Condition (formerly called Own State); Caregiver's Outlook; Quality of Care; Relationships; and Financial Worries. The total score is the mean of the 7 domain scores, with possible values ranging from 0 (worst possible quality of life) to 10 (best possible quality of life).

SECONDARY OUTCOMES:
Differences in trajectories of change between groups in McGill Quality of Life Questionnaire -Expanded [MQOL-E] domains | Trajectories over 12 months from start of enrollment in Stage 2 until study completion (assessments completed every two months))
  The McGill Quality of Life Questionnaire -Expanded has 20 items covering Physical, Psychological, Existential, Social, Feeling like a burden, Environment, Cognition and Quality of health care domains. Domain scores are calculated using the mean of the item scores assigned to each domain. Each domain has possible values ranging from 0 (worst possible) to 10 (best).
Differences in trajectories of change between groups in Quality of Life in Life-Threatening Illness- Family (version 3) domains | Trajectories over 12 months from start of enrollment in Stage 2 until study completion (assessments completed every two months))
  Quality of Life in Life-Threatening Illness- Family (version 3) includes 16 items measuring 7 domains that contribute to quality of life: Environment; Patient Condition; Caregiver's Own Condition (formerly called Own State); Caregiver's Outlook; Quality of Care; Relationships; and Financial Worries. Domain scores are calculated using the mean of the item scores assigned to each domain. Each domain has possible values ranging from 0 (worst possible) to 10 (best).
Differences in trajectories of change between groups in Canadian Health Care Evaluation Project Questionnaire [CANHELP] Lite Patient version Total Satisfaction Score | Trajectories over 12 months from start of enrollment in Stage 2 until study completion (assessments completed every two months))
  The patient version has 20 items and covers the following domains: Relationship with Doctors, Illness Management, Communication, Decision-Making, Your Well-being, and Overall Satisfaction. Three items on relationships with home health professionals adapted from the questions on relationships with doctors are added to the CANHELP-LITE assessment for patients to be used in this study. The Total Satisfaction score is the unweighted average of all answered questions. Each item has possible values ranging from 1 (worst possible) to 5 (best possible).
Differences in trajectories of change between groups in Canadian Health Care Evaluation Project Questionnaire [CANHELP] Lite Family version Total Satisfaction Score | Trajectories over 12 months from start of enrollment in Stage 2 until study completion (assessments completed every two months))
  The family caregiver version has 21 items representing the following domains: Relationship with Doctors, Characteristics of Doctors and Nurses, Illness Management, Communication and Decision-Making, Your Involvement, and Overall Satisfaction. Three items on relationships with home health professionals adapted from the questions on relationships with doctors are added to the CANHELP-LITE assessment for family caregivers to be used in this study. The Total Satisfaction score is the unweighted average of all answered questions. Each item has possible values ranging from 1 (worst possible) to 5 (best possible).
Differences in trajectories of change between groups in VR-12 (Veterans Rand 12) Physical Component Score (PCS) and a Mental Component Score (MCS). | Trajectories over 12 months from start of enrollment in Stage 2 until study completion (assessments completed every two months))
  VR-12 is a widely-used generic PROM which will be included for the measurement of general physical and mental health status and for cost-effectiveness analysis.
  VR-12 includes 12 original question items from the VR-36. The questions in this survey correspond to seven different health domains: general health perceptions, physical functioning, role limitations due to physical and emotional problems, bodily pain, energy/fatigue levels, social functioning and mental health. Answers are summarized into two scores, a Physical Component Score (PCS) and a Mental Component Score (MCS). Each question has possible values ranging from 1 (best possible) to 5 (worst possible).

CONTACTS AND LOCATIONS:
Overall Officials: Richard Sawatzky, Ph.D., Principal Investigator — Trinity Western University
Locations (2):
- Canada (2):
  - Alberta Health Services Edmonton Zone Home Living, Edmonton, British Columbia
  - BC Home Health Offices, Surrey, British Columbia

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data collected during the trial, after de-identification. Data will be shared through the Trinity Western University Dataverse site (currently under development). This includes all data obtained from patient and family caregiver completed quality of life and healthcare satisfaction questionnaires as well as economic evaluation questionnaires.
Supporting Information: Study Protocol, Analytic Code
Time Frame: Immediately following publication and up to 5 years after
Access Criteria: Anyone who wishes to access the data can do so through the Trinity Western University Dataverse (site currently under development - to be updated when link available). Data will be made available for any purpose.

REFERENCES:
- [Derived] Sawatzky R, Schick-Makaroff K, Ratner PA, Kwon JY, Whitehurst DGT, Ohlen J, Maybee A, Stajduhar K, Zetes-Zanatta L, Cohen SR. Did a digital quality of life (QOL) assessment and practice support system in home health care improve the QOL of older adults living with life-limiting conditions and of their family caregivers? A mixed-methods pragmatic randomized controlled trial. PLoS One. 2025 May 6;20(5):e0320306. doi: 10.1371/journal.pone.0320306. eCollection 2025. PMID 40327663